CLINICAL TRIAL: NCT05292820
Title: Exploring Sexual Function and Satisfaction of Trans Women After Vaginoplasty: Results of a Multicentric Survey
Brief Title: Sexual Function of Trans Women After Vaginoplasty
Acronym: GGAS-SEX
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0746
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Gender Dysphoria Vaginoplasty Sexuality
Keywords: Genital gender affirming surgery; Gender dysphoria; Transwomen; Vaginoplasty; Sexuality; Satisfaction
MeSH Terms: conditions — Gender Dysphoria; Sexuality; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transwomen vaginoplasty: Transgender women who underwent vaginoplasty
  Interventions: Other: Validated and non-validated questionnaire for exploration of sexuality and satisfaction after surgical procedure

INTERVENTIONS:
Other: Validated and non-validated questionnaire for exploration of sexuality and satisfaction after surgical procedure — Validated questionnaire : Female Sexual Function Index (FSFI), Female Genital Self-Imaging Scale (FGSIS), Body Image Scale (BIS), Non-validated questionnaire exploring post-surgery satisfaction, self-esteem scale, sexology.

SUMMARY:
Genital feminine affirming surgery may be an important step for transgender women. Vaginoplasty consists in the creation of external female genitalia and an operational vaginal cavity, and thus responds to major functional and aesthetic issues.

Different techniques are available: inversion of penile skin flap for creation of the vulva. The vaginal cavity may come from scrotal skin graft, sigmoid segment, small intestine, or peritoneal flap.

Vaginoplasty has a major place in the the transgender woman pathway, but the specific evaluation of long-term sexuality has not been explored so far.

Multicentric (Lyon, FR - Lille, FR - Limoges, FR), prospective, observational study Patients who underwent vaginoplasty or revision vaginoplasty.

Main objective:

To assess sexuality after sex reassignment surgery in transgender women.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Underwent vaginoplasty or revision in Lyon South Hospital, Lille University Hospital, Limoges University Hospital, between January 2007 and December 2019
* Penile inversion vaginoplasty with scrotal skin graft

Exclusion Criteria:

* < 18 years old
* Vaginoplasty other than scrotal skin graft : intestinal segment or peritoneal flap

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transwomen who underwent vaginoplasty or revision in Lyon, Lille, Limoges between January 2007 and December 2019
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
evaluation of FSFI : Female Sexual Function Index | At inclusion
  specific questionnaire scale
evaluation of FGSIS : Female Genital Self Imaging Scale | At inclusion
  specific questionnaire scale
evaluation of BIS : Body Image Scale | At inclusion
  specific questionnaire scale
evaluation of Rosenberg Self-esteem scale | At inclusion
  specific questionnaire scale

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Lille University Hospital, Lille
  - Limoges University Hospital, Limoges
  - Lyon South Hospital, Lyon

IPD SHARING:
Plan to Share IPD: Undecided